CLINICAL TRIAL: NCT05844761
Title: Real-time Motion Management During Prostate and Lung Radiotherapy
Acronym: REMIND
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, André Änghede Haraldsson, Principal Investigator, Region Skane
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-05273-01
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cancer of Lung; Lung Metastasis; Cancer of Prostate
MeSH Terms: conditions — Lung Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will undergo radiotherapy using motion management techniques: Triggered Imaging with TrueBeam for prostate cancer, Synchrony with Radixact for prostate cancer, and Synchrony with Radixact for lung cancer. Dosimetric coverage will be assessed after treatment based on the accuracy of the motion management techniques and compared with dose coverage without motion management. After interim analysis, Planning target volume (PTV) will be reduced based on dosimetric accuracy in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Triggered Imaging with TrueBeam for prostate cancer (Experimental): Patients will undergo radiotherapy using the Triggered Imaging technique with TrueBeam for prostate cancer. The technology on the TrueBeam allows for monitoring and gating of the radiation beam in relation to the target position.
  Interventions: Radiation: Triggered imaging on TrueBeam with margin reduction
- Synchrony with Radixact for prostate cancer (Experimental): Patients will undergo radiotherapy using the Synchrony technique with Radixact for prostate cancer. Multi-Leaf Collimator Adaptation (MLC) and kilovoltage (kV) Intrafraction Monitoring with the Synchrony technique on the Radixact radiotherapy machine.
  Interventions: Radiation: Synchrony MLC tracking on fiducials with margin reduction
- Synchrony with Radixact for lung cancer (Experimental): Patients will undergo radiotherapy using the Synchrony technique with Radixact for lung cancer. MLC Adaptation, Respiratory Motion Tracking, and kV Intrafraction Monitoring with the adaptive Synchrony technique on the Radixact radiotherapy machine.
  Interventions: Radiation: Synchrony MLC tracking and lung adaptive model with margin reduction

INTERVENTIONS:
Radiation: Triggered imaging on TrueBeam with margin reduction — At interim analysis the Planning target volume (PTV) will be reduced based on the accuracy of the TrueBeam triggered imaging motion management technique.
  Arms: Triggered Imaging with TrueBeam for prostate cancer
Radiation: Synchrony MLC tracking on fiducials with margin reduction — At interim analysis the Planning target volume (PTV) will be reduced based on the accuracy of the Radixact Synchrony motion management technique.
  Arms: Synchrony with Radixact for prostate cancer
Radiation: Synchrony MLC tracking and lung adaptive model with margin reduction — At interim analysis the Planning target volume (PTV) will be reduced based on the accuracy of the Radixact Synchrony motion management technique for lung cancer.
  Arms: Synchrony with Radixact for lung cancer

SUMMARY:
The goal of this interventional non-inferiority trial is to assess the accuracy of different real-time motion management radiotherapy techniques. The main question the study aims to answer are:

* What are the target margins for radiotherapy with motion management that are not inferior to target margin without motion management
* What are the dosimetric and geometrical accuracy to patient for the motion management techniques.

Participants will answer QoL questionary, and the accuracy of treatment will be assessed from treatment data.

DETAILED DESCRIPTION:
This study will assess the feasibility of implementing real-time tracking in a clinical setting to account for the relative motion of the moving tumours localised to the prostate or lung. The capability to track the treatment target's motion will ensure that the dose prescribed by the radiation oncologist is the dose delivered to the target and minimises side effects to the critical organs.

During radiation treatment, the target position will be monitored in real-time using built-in imaging technology. The radiation beam shape will be altered to compensate for the moved target positions by the treatment delivery system. The delivered dose to the patient will be calculated after the treatment and compared to the dose without real-time tracking to assess the potential benefit to treatment efficacy, recognising that the radiation dose received by tumour tissue is a very strong biomarker for response.

The estimated dose distributions will be compared to the original plan for non-inferiority using the dose reconstruction method based on the prostate motion trajectory and the logged MLC positions (beam shapes).

Also, the impact on organs at risk doses due to MLC target tracking.

ELIGIBILITY:
Inclusion Criteria:

For prostate cancer patients:

* Patients histologically proven prostate adenocarcinoma
* Prostate specific antigen (PSA) obtained within three months prior to enrollment
* Localised prostate cancer at any stage eligible for radiotherapy: i.e. any T- or Gleason stage, but no pelvic lymph nodes can be included within the target to be treated
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document.
* Hypofractionated radiation therapy (HYPO) fractionated patients with a prescribed dose of 42.7Gy in 7 fractions.
* MRIOnly workflow meaning synthetic generated CT based on Magnetic resonance imaging (MRI)
* Patients over 40 years old

For lung cancer patients:

* Lung cancer or localised metastatic disease from other cancer diagnoses, accepted for stereotactic radiotherapy to 45Gy in 3 fractions
* Lesion distinguishable on Computer Tomography and where the majority of adjacent tissue is the lung.
* Ability to understand and the willingness to sign a written informed consent document.
* Is able to perform treatment simulation

Exclusion Criteria:

For prostate cancer patients:

* Patient must have three gold fiducial markers inserted in the prostate
* Patients with artificial Hip(s), lumbar spinal surgical rods or other large metallic pelvic implants
* Patients with overlapping implanted gold fiducials in X-ray imaging
* Unfeasible to track fiducials with kv imaging/existing online imaging systems

For lung cancer patients:

* Previous treatment with radiotherapy for lung cancer or lung metastasis
* Idiopathic lung fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dosemetric accuracy | At treatment completion, approximately 1-4 weeks
  Dose coverage defined as dose to 99% of clinical target volume (CTV) (D99%) to target including margin for other uncertainties.

SECONDARY OUTCOMES:
Geometric accuracy | At treatment completion, approximately 1-4 weeks
  The geometric accuracy of the beam shape, determined by comparing the ideal beam shape with the actual beam shape based on the centroid of the shape as assessed with mean absolute error (MAE)
Motion trajectory | At treatment completion, approximately 1-4 weeks
  Motion trajectory measured by kilovoltage imaging, including any prediction algorithms compared to without latency and other limitations compared with MAE.
Acute Toxicity | Baseline prior to first fraction. At end of radiotherapy (1-4 weeks) and at 3 months after last fraction..
  EORTC guided and physician assessed
Mechanical & software failure | At treatment completion, approximately 1-4 weeks
  The percentage of fractions delivered without software or mechanical failure

CONTACTS AND LOCATIONS:
Overall Officials: André Haraldsson, PhD, MPE, Principal Investigator — Skane university hospital, Lund university
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data used in this study contains sensitive information about the study participants and they did not provide consent for public data sharing. The current approval by the Swedish Ethical Review Authority does not include data sharing. A minimal data set could be shared by request from a qualified academic investigator for the sole purpose of replicating the present study, provided the data transfer is in agreement with European Union legislation on the general data protection regulation and approval by the Swedish Ethical Review Authority.
Supporting Information: Study Protocol
Time Frame: <1y after study. At least 5 years
Access Criteria: On request and as supplementary at publication